CLINICAL TRIAL: NCT04726761
Title: Frequent Cuff Inflations May Disrupt the Accuracy of 24-hour Ambulatory Blood Pressure Monitoring
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 1337
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
Keywords: Ambulatory Blood Pressure Monitoring; ABPM
MeSH Terms: conditions — Hypertension | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frequent/Non-frequent: Patients randomized to this order will first have an ABPM conducted with the frequent measuring intervals (3 times an hour during day and 2 times an hour at night) and then a few days later have another ABPM conducted with the non-frequent measuring interval (1 time an hour during all 24 hours)
  Interventions: Diagnostic Test: Ambulatory Blood Pressure Monitoring, frequent/non-frequent
- Non-frequent/frequent: Patients randomized to this order will first have an ABPM conducted with the non-frequent measuring interval (1 time an hour during all 24 hours) and then a few days later have another ABPM conducted with the frequent measuring intervals (3 times an hour during day and 2 times an hour at night)
  Interventions: Diagnostic Test: Ambulatory Blood Pressure Monitoring, non-frequent/frequent

INTERVENTIONS:
Diagnostic Test: Ambulatory Blood Pressure Monitoring, frequent/non-frequent — Patient will have a Spacelabs 90217 attached. This device can automatically measure the blood pressure over 24 hours. Patients will have their blood pressure measured first with a frequent interval, and then a non-frequent interval.
  Groups: Frequent/Non-frequent
Diagnostic Test: Ambulatory Blood Pressure Monitoring, non-frequent/frequent — Patient will have a Spacelabs 90217 attached. This device can automatically measure the blood pressure over 24 hours. Patients will have their blood pressure measured first with a non-frequent interval, and then a frequent interval.
  Groups: Non-frequent/frequent

SUMMARY:
24-hour ambulatory blood pressure monitoring (ABPM) is superior to office blood pressure (BP) for assessing cardiovascular risk. On the other hand, repeated cuff inflations during ABPM can cause discomfort and reduced quality of sleep. A high frequency of measurement during ABPM might result in erroneously high BP measurement, incorrect hypertension diagnoses, unnecessary treatment or just overtreatment with antihypertensive medication and potentially serious side effects.

The purpose of this study is to investigate whether the frequency of measurements during ABPM impacts the measured BP during ABPM.

Patients will be recruited from the Clinic of Hypertension at Aarhus University Hospital, Denmark. The study will be conducted as a randomized controlled crossover study. Participants will undergo two 24-hour ABPMs: One with a low frequency of measurement, 1-time per hour during the day and 1-time per hour during the night, and one with a high frequency, 3-times/hour during the day, and 2-times/hour at night. The primary endpoint will be the difference in 24-hour mean systolic BP between the high- and low frequency measurement ABPM.

DETAILED DESCRIPTION:
Aim:

The purpose of this study is to evaluate if 24-hour ABPM with frequent BP measurements (intervals of 20 minutes during daytime and 30 minutes during nighttime) result in erroneously elevated BP in hypertensive patients compared with non-frequent BP readings (measurement intervals of 60 minutes both day and night).

Population:

The study population will comprise all patients referred to and attending the Clinic of Hypertension, AUH, who are scheduled to undergo ABPM. At referral to the Clinic of Hypertension, AUH, patients will be contacted with an electronic or analog letter, informing them about the study and inviting them to participate. Patients who already are being treated at the Clinic of Hypertension, will be invited at an appointment in the clinic. Patients will be excluded from the study if they have atrial fibrillation, nighttime work, insomnia or sleeping disorders, and are not physically able to undergo an ABPM (e.g. too big arm circumference to fit the cuff).

Methods:

This will be a randomized controlled crossover study (figure 2). At arrival patients will be fitted with the device, a SPACELABS 90217 by a nurse. The nurse will conduct an office blood pressure measurement, in accordance with ESH guidelines to be sure the device is working, and for later comparison. Patients will have their first ABPM conducted with either frequent or non-frequent ABPM measurement protocol as described above, randomized 1:1. Patients will be instructed to remove their device after 24 hours of measurement and have an appointment to return the device between 2-7 days. At least two days between measurements ensure a sufficient washout period. The maximum of 7 days before second measurement makes sure the patient's appointment with a doctor at the clinic will not be delayed. When returning the device, patients will have the same device mounted again, measuring with the frequency not assigned at the initial randomization. Participants will be instructed to repeat the same procedures regarding the device and to, as far as possible, conduct the same daily activities on the second day of measurement as during the first day of measurement. Patients will not have any alterations in blood pressure medication between the two measuring days. After each ABPM, patients will answer a routine questionnaire from the clinic about sleep, discomfort, pain, and the degree to which the device caused interference with daily activities and/or disturbance of sleep. Since the questionnaire is standard procedure at the clinic, we will be able to compare characteristics between the group who are not interested in joining the study and patients do participate. In this way the investigators can ensure no unknown selection bias occurs. Both ABPM will be used by the clinician at the appointment in the clinic.

Sample size:

In a pilot study conducted at the Clinic of Hypertension, AUH, the investigators found a mean difference of 7 mmHg (Standard deviation = 13,76) between a 20-minute interval and a 1-hour interval between measurements, respectively. Using a sample size calculation, for crossover design with quantitative measurement, a two-sided significance level of 0.025 and a power of 0.9, and a minimal clinical difference of 10mmHg, we calculate a minimum sample size of 38 patients. It is estimated only 25% of patients with this difference will be in intermediate hypertension group as studied in the previous pilot study, which is why 152 patients wil be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients either has to be referred from primary care to the Clinic of Hypertension at Aarhus University hospital, or already being treated at the clinic. Both groups has to be scheduled for a 24-hour ambulatory blood pressure monitoring.

Exclusion Criteria:

* Below 18 years of age
* Have atrial fibrillation
* Have routine nightshift work
* Is pregnant
* Is physically inable to have the cuff applied correctly (too large arm circumference)
* Known insomnia or other sleeping disorders
* Change in blood pressure medication within 14 days before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients, either referred or existing patients, who has to undergo a 24-hour ambulatory blood pressure monitoring
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
The difference in mean systolic blood pressure (SBP) between 24-hour ABPM with frequent and non-frequent measurement intervals | One week
  The systolic blood pressure is one of the most important predictors of a patient's risk of cardiovascular disease that can be measured with ABPM.

SECONDARY OUTCOMES:
The difference in mean diastolic blood pressure (DBP) between 24-hour ABPM with frequent and non-frequent measurement intervals. | One week
  Diastolic blood pressure is an important predictor of a patient´s risk of cardiovascular disease that can be measured with ABPM.
The self-reported pain/discomfort, interference in daily life, and disturbance of sleep during frequent and non-frequent measurement ABPM | One week
  Self-reported data from a questionnaire, to see if there is a correlation between these factors and a possible difference in measured blood pressure.
The difference in average real variability (ARV), dipping status and morning surge during frequent and non-frequent measurement ABPM. | One week
  These are less common but also important factors in regards of a patients blood pressure profile, used to asses a patient's risk of cardiovascular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Henrik Buus, Study Chair — Klinisk Institut, Aarhus Universitets Hospital
Locations (1):
- Hypertension Clinic, Aarhus University Hospital, Aarhus, Denmark